CLINICAL TRIAL: NCT00579046
Title: Erythropoietin Treatment of Anemia Complicating Chronic Obstructive Pulmonary Disease: Functional Impact During Exertion
Brief Title: Study of Erythropoietin to Treat Anemia Complicating Chronic Obstructive Pulmonary Disease
Acronym: ELAB
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: no patient recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 061011
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Anemia; Chronic Obstructive Pulmonary Disease
Keywords: Anemia; Chronic obstructive Pulmonary Disease; Erythropoietin; 6-minute walk test
MeSH Terms: conditions — Anemia; Pulmonary Disease, Chronic Obstructive | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — Dosage form: injection (to store between 2 and 8 °C). Dosage: various dosages are available (10, 15, 20, 30, 40, 50, 60, 80, 100, 150 or 300 µg/ml).
  Frequency: every week for 2 months: 8 injections

SUMMARY:
The purpose of this study is to determine the impact of erythropoietin treatment of anemia on exercise capacity of patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The development of anemia in patients with chronic obstructive pulmonary disease (COPD) is now taken as a predictor of increased morbidity and mortality. Preliminary data from patients investigated in our department indicate a negative correlation between anemia severity and 6-minute walking distance. Our working hypothesis is that hemoglobin level correction by erythropoietin therapy will improve the effort capacity of patients with COPD and anemia. Our objective is to conduct a pilot study of the efficacy of darbepoetin alfa.

The study will include about 15 patients with COPD recruited at three pulmonology centers based on two selection criteria: COPD stage II or III or IV according to GOLD criteria and hemoglobin level less than 12 g/dL. Effort capacity will be evaluated chiefly by performing a 6-minute walking test and by measuring VO2 at maximum exertion on a bicycle ergometer with increasing loads. Darbepoetin alfa will be given for 2 months. If the hemoglobin increase is less than 1 g/dL after 1 month, the dosage will be increased by 25%.

Effort parameters will be measured at baseline and after 1 and 2 months of treatment. Among secondary objectives, we will evaluate functional ergospirometric parameters and laboratory tests for inflammation. Total study duration will not exceed 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 40-75 years
* Diagnosis of a moderate to very severe COPD (stage II, III or IV according to GOLD criteria)
* A ratio of post-bronchodilator FEV1 to forced vital capacity (FVC) < 70%
* A FEV1 < 80% of the predicted value
* Hemoglobin level less than 12 g/dL
* Peak VO2 less than 80% of predict value and 6-min walk test distance less than 500 meters

Exclusion Criteria:

* Hemorrhagic anemia
* Iron deficiency anemia (ferritin < 30 ng/ml)
* Folate and Vitamin B12 deficiency anemia
* Myelodysplastic Syndrome
* Chronic disease associated with anemia: renal insufficiency, inflammatory disease, neoplastic disease, left ventricular insufficiency (ejection fraction < 40%)
* Chronic disease likely to interfere with dyspnea or exercise testing (cardiac insufficiency, neurologic disease, claudication)
* Acute exacerbation of COPD within the last 4 weeks
* History of thromboembolic disease
* Contraindications for cardiopulmonary exercise testing
* Contraindications for darbepoetin alfa treatment: uncontrolled arterial hypertension or hypersensitivity reaction to darbepoetin alfa
* Pregnancy or breast-feeding (women of reproductive potential should use adequate birth control measures during the whole duration of study treatment)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Measure: 6-minute walk distance | before treatment; at one month and two months of treatment

SECONDARY OUTCOMES:
VO2 max | before treatment; at one month and two months
MRC Dyspnea score | before treatment; at one month and two months
St. George quality of life score | before treatment and at two months of treatment
Inflammation biological parameters | before treatment and at two months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Savale, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France